CLINICAL TRIAL: NCT05633212
Title: Binocular Vision Alternations and Functional Magnetic Resonance Imaging Activation After Implantable Collamer Lens Implantation for High Myopia
Brief Title: Binocular Vision Alternations and fMRI Activation After ICL Implantation for High Myopia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Other Study IDs: 2022KYPJ198
Record Dates: First submitted 2022-11-03; First posted 2022-12-01 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-03

CONDITIONS: Binocular Vision Disorder
Keywords: binocular vision, accommodation, vergence, fMRI

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Implantable collamer lens (ICL) is one of the most effective operation for high myopia. Due to refractive correction changed, and prism effect of the spectacle removed, in the early stage after ICL implantation, binocular function might be dysfunction, leading to asthenopia, blurred vision, double vision and so on. This study will recruit the high myopia subjects that scheduled for ICL implantation, purpose to investigate the binocular vision alternations and brain activation that impacted by ICL implantation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-35
* Spherical equivalent over -6.00DS, astigmatism within -2.00DC, anisometropia within -2.00DS
* BCVA ≥ 0.8
* Plan to accept implantable collamer lens surgery
* Near point of convergence within 10cm
* Positive fusion vergence over 20pd

Exclusion Criteria:

* Stabismus
* Previous ocular surgery or trauma
* History of vision therapy
* Monovision and nystagmus
* Mental disease or craniocerebral trauma

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The high myopia subjects that scheduled for ICL implantation from Zhongshan Ophthalmic Center, Sun Yat-sen University
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of phoria at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Phoria was measured by phoropter.
Changes of AC/A at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Gradient AC/A was measured by phoropter.
Changes of fusion vergence at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Fusion vergence was measured by phoropter.
Changes of accommodative response at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Accommodative response was measured using monocular estimated method.
Changes of relative accommodation at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Relative accommodation was measured by phoropter.
Changes of near point of convergence at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Near point of convergence was measured using push-up method.
Changes of accommodation amplitude at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Accommodative amplitude was measured using push-up method.
Changes of vergence facility at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Vergence facility was measured by +2.00D/-2.00D flipper.
Changes of accommodative facility at different time points | The examination was performed before operation and 1 week, 1 month, 3 monthes, 6 monthes after ICL implantation.
  Accommodative facility was measured by 3△BI/12△BO flipper.

SECONDARY OUTCOMES:
Changes of brain activation at different time points | The examination was performed before operation and 1 month, 6 monthes after ICL implantation.
  Functional magnetic resonance imaging activation of the brain

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zheng K, Han T, Zhou X. Accommodative changes after SMILE for moderate to high myopia correction. BMC Ophthalmol. 2016 Oct 4;16(1):173. doi: 10.1186/s12886-016-0352-8. PMID 27716112
- [Background] Han J, Hong S, Lee S, Kim JK, Lee HK, Han SH. Changes in fusional vergence amplitudes after laser refractive surgery for moderate myopia. J Cataract Refract Surg. 2014 Oct;40(10):1670-5. doi: 10.1016/j.jcrs.2014.01.043. Epub 2014 Aug 20. PMID 25149555
- [Background] Tsujimoto K, Mizuno K, Nishida D, Tahara M, Yamada E, Shindo S, Kasuga S, Liu M. Prism adaptation changes resting-state functional connectivity in the dorsal stream of visual attention networks in healthy adults: A fMRI study. Cortex. 2019 Oct;119:594-605. doi: 10.1016/j.cortex.2018.10.018. Epub 2018 Oct 31. PMID 30471844
- [Background] Wilf M, Serino A, Clarke S, Crottaz-Herbette S. Prism adaptation enhances decoupling between the default mode network and the attentional networks. Neuroimage. 2019 Oct 15;200:210-220. doi: 10.1016/j.neuroimage.2019.06.050. Epub 2019 Jun 22. PMID 31233909
- See also: Accommodative changes after SMILE for moderate to high myopia correction. — https://pubmed.ncbi.nlm.nih.gov/27716112/
- See also: Changes in fusional vergence amplitudes after laser refractive surgery for moderate myopia. — https://pubmed.ncbi.nlm.nih.gov/25149555/
- See also: Prism adaptation changes resting-state functional connectivity in the dorsal stream of visual attention networks in healthy adults: A fMRI study. — https://pubmed.ncbi.nlm.nih.gov/30471844/
- See also: Prism adaptation enhances decoupling between the default mode network and the attentional networks. — https://pubmed.ncbi.nlm.nih.gov/31233909/